CLINICAL TRIAL: NCT03568435
Title: Efficacy and Safety of Nivolumab in Metastatic Renal Cell Cancer Patients - Japanese Real-World Data Through Clinical Chart Review
Brief Title: Safety and Effectiveness of Nivolumab in Recurring Kidney Cancer Participants
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-8D3
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Kidney Cancer; Renal Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with metastatic RCC taking nivolumab: Specified dose on specified day
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
A non-interventional, medical record review of clinical data collected from Japanese participants with recurring kidney cancer

ELIGIBILITY:
Inclusion Criteria:

* A patient with RCC with distant metastasis treated for the first time with nivolumab

Exclusion Criteria:

* Patients who have participated in some trials with immuno-checkpoint blockade before or after treatment with nivolumab after diagnosis with RCC

Other protocol defined inclusion/exclusion criteria could apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with RCC with distant metastasis treated with nivolumab under real clinical practice
Sampling Method: Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Overall survival status | 6 months
Overall survival status | 36 months
Best overall response | 6 months
Best overall response | 36 months
Progression free survival rate | 6 months
Progression free survival rate | 36 months
Disease free survival | 6 months
Disease free survival | 36 months
Objective response rate | 6 months
Objective response rate | 36 months
Duration of response | 6 months
Duration of response | 36 months
Incidence of adverse events | 36 months
Incidence of serious adverse events | 36 months

SECONDARY OUTCOMES:
Distribution of clinical characteristics | 36 months
Distribution of socio-demographic characteristics | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm